CLINICAL TRIAL: NCT06839560
Title: A Prospective, Multicenter, Randomized Controlled Phase II Study to Evaluate the Efficacy and Safety of PD-L1 Monoclonal Antibody Combined with VEX Metronomic Chemotherapy and Concurrent or Delayed Radiotherapy in Patients with Advanced HER2-Negative Breast Cancer with Brain Metastasis
Brief Title: Evaluating the Efficacy and Safety of PD-L1 Monoclonal Antibody Combined with VEX Metronomic Chemotherapy and Concurrent or Delayed Radiotherapy in Patients with Advanced HER2-Negative Breast Cancer with Brain Metastasis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ma Fei，MD, Deputy Director of the Department of Medical Oncology, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC5108
Record Dates: First submitted 2025-02-18; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2024-09

CONDITIONS: Brain Metastasis from Advanced HER2-negative Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Concurrent Radiotherapy) (Experimental): 1. Adelumab: 1200 mg on Day 1, every 3 weeks (q3w).
  2. VEX Metronomic Chemotherapy:
  1) Vinorelbine: 20 mg orally, every other day, every 3 weeks (q3w). 2) Cyclophosphamide: 50 mg orally, once daily, every 3 weeks (q3w). 3) Capecitabine: 500 mg orally, three times daily, every 3 weeks (q3w). 3. Radiotherapy: The interval between radiotherapy and immunotherapy should be within 3 weeks, with no specific order required. Different radiotherapy techniques will be selected based on the size and location of the metastatic lesions:
  1. Stereotactic Body Radiation Therapy (SBRT),
  2. Spatially Fractionated Radiation Therapy (SFRT),
  3. Low-dose Radiotherapy (LDRT).
  Interventions: Drug: Adelumab+VEX Metronomic Chemotherapy+Concurrent Radiotherapy
- Control Group (Delayed Radiotherapy) (Active Comparator): 1. Adelumab: 1200 mg on Day 1, every 3 weeks (q3w).
  2. VEX Metronomic Chemotherapy:
  1) Vinorelbine: 20 mg orally, every other day, every 3 weeks (q3w). 2) Cyclophosphamide: 50 mg orally, once daily, every 3 weeks (q3w). Capecitabine: 500 mg orally, three times daily, every 3 weeks (q3w). 3. Radiotherapy: If there is intracranial disease progression but extracranial disease remains stable, the systemic treatment regimen of Adelumab + VEX metronomic chemotherapy will be continued, with the addition of intracranial radiotherapy.
  If there is intracranial disease progression and extracranial disease progression, the systemic treatment regimen will be modified, with the addition of intracranial radiotherapy. The radiotherapy positioning and techniques will be the same as those used in the experimental group.
  Interventions: Drug: Adelumab+VEX Metronomic Chemotherapy+Delayed Radiotherapy

INTERVENTIONS:
Drug: Adelumab+VEX Metronomic Chemotherapy+Concurrent Radiotherapy — 1. Adelumab: 1200 mg on Day 1, every 3 weeks (q3w).
  2. VEX Metronomic Chemotherapy:
     Vinorelbine: 20 mg orally, every other day, every 3 weeks (q3w). Cyclophosphamide: 50 mg orally, once daily, every 3 weeks (q3w). Capecitabine: 500 mg orally, three times daily, every 3 weeks (q3w).
  3. Radiotherapy: The interval between radiotherapy and immunotherapy should be within 3 weeks, with no specific order required. Different radiotherapy techniques will be selected based on the size and location of the metastatic lesions:
  Stereotactic Body Radiation Therapy (SBRT), Spatially Fractionated Radiation Therapy (SFRT), Low-dose Radiotherapy (LDRT).
  Arms: Experimental Group (Concurrent Radiotherapy)
Drug: Adelumab+VEX Metronomic Chemotherapy+Delayed Radiotherapy — 1. Adelumab: 1200 mg on Day 1, every 3 weeks (q3w).
  2. VEX Metronomic Chemotherapy:
     Vinorelbine: 20 mg orally, every other day, every 3 weeks (q3w). Cyclophosphamide: 50 mg orally, once daily, every 3 weeks (q3w). Capecitabine: 500 mg orally, three times daily, every 3 weeks (q3w).
  3. Radiotherapy:
  If there is intracranial disease progression but extracranial disease remains stable, the systemic treatment regimen of Adelumab + VEX metronomic chemotherapy will be continued, with the addition of intracranial radiotherapy.
  If there is intracranial disease progression and extracranial disease progression, the systemic treatment regimen will be modified, with the addition of intracranial radiotherapy.
  The radiotherapy positioning and techniques will be the same as those used in the experimental group.
  Arms: Control Group (Delayed Radiotherapy)

SUMMARY:
A Prospective, multicenter, randomized controlled phase II study to evaluate the efficacy and safety of PD-L1 monoclonal antibody combined with vinorelbine + cyclophosphamide + capecitabine (VEX) metronomic chemotherapy and concurrent or delayed radiotherapy in patients with advanced HER2-negative breast cancer with brain metastasis

ELIGIBILITY:
Inclusion Criteria:

1. Males or females who are at least 18 years of age on the day of signing the informed consent form.
2. Patients with metastatic HER2-negative breast cancer brain metastasis, with clear clinical documentation; specific criteria refer to the guidelines of the American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP).
3. Patients who have received no more than one line of chemotherapy during the metastatic stage of breast cancer.
4. Patients with brain metastasis should not require immediate local therapy during the trial and meet at least one of the following criteria:

   1. The patient has not previously received intracranial radiotherapy.
   2. The patient has not previously undergone surgery for intracranial metastases; if surgery was performed, the surgical lesion is not the target for the planned radiotherapy, or it is the target lesion and has recurred after surgery.
5. The patient must have at least one measurable intracranial lesion, with the longest diameter baseline accurately measurable by magnetic resonance imaging (MRI) as ≥10 mm and suitable for precise repeated measurement according to RECIST 1.1 in combination with RANO criteria. Measurable extracranial lesions are not required.
6. Patients with suspected or confirmed leptomeningeal metastasis should be excluded.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1, assessed within 10 days before the start of study treatment.
8. Patients may have previously received anthracycline (e.g., doxorubicin, epirubicin) and/or taxane (e.g., paclitaxel, docetaxel) therapy, specifically including:

   1. Before breast cancer recurrence, the patient received anthracycline and/or taxane during adjuvant or neoadjuvant treatment.
   2. The patient experienced treatment failure during or after anthracycline and/or taxane-based chemotherapy.
   3. In the judgment of the investigator, the patient is not suitable for anthracycline and/or taxane-based chemotherapy as a first-line treatment regimen.
9. Female patients are not pregnant, not breastfeeding, and agree to use necessary contraceptive measures.
10. The patient is able to sign the informed consent form to participate in the study.
11. The patient has adequate organ function, as detailed in Table 1 of the study protocol; all screening laboratory tests should be completed within 10 days before the start of study treatment.

Exclusion Criteria:

1. The subject has leptomeningeal metastasis.
2. If the patient has concurrent brain metastasis, the neurological symptoms are too severe to cooperate with radiotherapy.
3. Malabsorption syndrome, or the disease significantly affects gastrointestinal function; or after subtotal gastrectomy, or after proximal small bowel resection, which may affect the absorption of oral metronomic chemotherapy agents.
4. The subject has dysphagia or is unable to swallow tablets.
5. Known history of another invasive malignancy that is progressing or requires active treatment within the past 5 years. (Subjects with a history of cutaneous basal cell carcinoma, squamous cell carcinoma of the skin, ductal carcinoma in situ of the breast treated with curative intent, or in situ cervical cancer are not excluded.)
6. Previous treatment with anti-PD-1, anti-PD-L1, or anti-PD-L2 agents, or targeted drugs acting on another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX40, CD137).
7. Diagnosis of immunodeficiency or receiving long-term systemic corticosteroid therapy (daily dose exceeding 10 mg prednisone equivalent) or any form of immunosuppressive therapy within 7 days before the first dose of study treatment.
8. Active autoimmune disease requiring systemic treatment within the past 2 years (e.g., use of disease-modifying drugs, corticosteroids, or immunosuppressive agents).
9. History of pneumonia requiring steroid treatment (non-infectious) or current pneumonia.
10. Positive urine pregnancy test within 72 hours before the first dose of study treatment.
11. Active infection requiring systemic treatment.
12. Known history of active tuberculosis.
13. Echocardiogram performed at screening confirms left ventricular ejection fraction (LVEF) <50% or below the institutional lower limit of normal.
14. Other significant cardiac disease, such as: myocardial infarction, acute coronary syndrome, or history of coronary artery angioplasty/stent placement/bypass surgery within the past 6 months; New York Heart Association (NYHA) Class II-IV congestive heart failure (CHF) or history of NYHA Class III or IV CHF.
15. Known history of human immunodeficiency virus (HIV) infection.
16. Known history of hepatitis B (defined as positive hepatitis B surface antigen [HBsAg]) or known active hepatitis C virus infection (defined as detectable HCV RNA [qualitative]).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2028-09-10 (Estimated); Study Completion 2028-09-10 (Estimated)

PRIMARY OUTCOMES:
Intracranial Progression-Free Survival (iPFS) | 24 months
  According to RECIST 1.1 criteria：Disease Progression (PD): Referring to the smallest sum of the diameters of all measured target lesions throughout the entire experimental study, there is a relative increase of at least 20% in the sum of the diameters (if the baseline measurement is the smallest, then the baseline value is used as the reference); in addition, there must be an absolute increase of at least 5 mm in the sum of the diameters (the appearance of one or more new lesions is also considered disease progression).

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing 100021, Beijing, Beijing Municipality, China